CLINICAL TRIAL: NCT06857552
Title: The Effect of Ultrasound Guided Visual Biofeedback Performed by Midwifes on the Duration of the Active Second Stage of Labor, a Randomized Controlled Trial
Brief Title: The Effect of Ultrasound Guided Visual Biofeedback Performed by Midwifes on the Duration of the Active Second Stage of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaplan Medical Center (Other)
Responsible Party: Principal Investigator, Roni Levy, Head of Labor and Delivery, Kaplan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0029-21-KMC
Record Dates: First submitted 2025-02-23; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Labor Stage, Second
Keywords: Prolonged second stage; Transperineal ultrasound; biofeedback
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Coached maternal pushing via ultrasound (US) (Experimental): The study group, will have coached pushing using trans-perinal ultrasound (US) performed by the midwife during the active stage of labor, and after diagnosis of complete dilatation. Further, if not delivered within 2 hours of complete dilatation, a third coaching will be conducted. The coaching process in each will be performed for 10 minutes and for at least 3 contractions.
  In the study group the women will observe the fetal head movements on the screen in front of her.
  Interventions: Other: Visual biofeedback using transperineal ultrasound (TPUS)
- Traditional coached maternal pushing (No Intervention): The control group will have the traditional coached pushing (vaginal) performed by a midwide during the active stage of labor, and after diagnosis of complete dilatation. Further, if not delivered within 2 hours of complete dilatation, a third coaching will be conducted. The coaching process in each will be performed for 10 minutes and for at least 3 contractions The women in the controlled group will have the vocal coaching of the midwife during the contractions.

INTERVENTIONS:
Other: Visual biofeedback using transperineal ultrasound (TPUS) — The intervention (study) arm will recieve coached maternal pushing via transperineal ultrasound (US) with visual biofeedback
  Arms: Coached maternal pushing via ultrasound (US)

SUMMARY:
The goal of this randomized controlled trial is to investigate whether using of coached sonographic pushing will decrease the length of the second stage of labor and the rate of operative deliveries.

Researchers will compare women who undergo the traditional coached pushing to women who undergo visual biofeedback coached pushing.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Nulliparous
* 37-42 weeks of gestation
* Under neuroaxial analgesia
* Reached the second stage of labor
* An estimated fetal weight between 2500-4000 grams

Exclusion Criteria:

* Women who arrived in active labor and delivered before being assessed by a physician.
* Women with contra-indications for vaginal birth

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2024-09-07 (Actual)

PRIMARY OUTCOMES:
Length of the second stage of labor | At baseline
  To investigate whether using of coached sonographic pushing will decrease the length of the second stage of labor.
Mode of delivery | At baseline
  To investigate whether using of coached sonographic pushing will affect the rate of operative deliveries.

SECONDARY OUTCOMES:
Maternal outcomes | At baseline
  Maternal 3rd or 4th degree tear rate, postpartum hemorrhage rates
Neonatal Outcomes | At baseline
  Neonatal cord PH
Neonatal Outcomes | At baseline
  Apgar score less than 7 in 5 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaplan Medical Center, Rehovot, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bellussi F, Alcamisi L, Guizzardi G, Parma D, Pilu G. Traditionally vs sonographically coached pushing in second stage of labor: a pilot randomized controlled trial. Ultrasound Obstet Gynecol. 2018 Jul;52(1):87-90. doi: 10.1002/uog.19044. Epub 2018 May 30. PMID 29532533
- [Background] Gilboa Y, Frenkel TI, Schlesinger Y, Rousseau S, Hamiel D, Achiron R, Perlman S. Visual biofeedback using transperineal ultrasound in second stage of labor. Ultrasound Obstet Gynecol. 2018 Jul;52(1):91-96. doi: 10.1002/uog.18962. Epub 2018 May 29. PMID 29155474